CLINICAL TRIAL: NCT01012635
Title: Cortical Modulation of Chronic Pain
Brief Title: Chronic Pain and Brain Activity in Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Mark Jensen, Professor, University of Washington
Other Study IDs: 36127-B; 1R21HD058049-01A2 (NIH)
Record Dates: First submitted 2009-10-30; First posted 2009-11-13 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; chronic pain
MeSH Terms: conditions — Spinal Cord Injuries; Chronic Pain | interventions — Hypnosis; Meditation; Biofeedback, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Neurofeedback, tDCS (2 levels), Self-hypnosis, Meditation
  Interventions: Other: Hypnosis; Other: Meditation; Other: Neurofeedback training; Other: Two different levels of tDCS

INTERVENTIONS:
Other: Hypnosis — Hypnosis Training: Verbal suggestions from an audio recording (via headphones).
Other: Meditation — Meditation: focus on a single word ("one") for the entire session.
Other: Neurofeedback training — Neurofeedback Training: Two electrodes will be placed on your scalp, and one electrode clipped on your head. There is no risk of electrical shock.
  Other Names: biofeedback
Other: Two different levels of tDCS — Direct stimulation of the brain by using a weak electrical current. There is no risk of electrical shock.

SUMMARY:
This study compares five different procedures to see how they affect pain and brain activity. The procedures include neurofeedback, self-hypnosis training, meditation, and two different levels of transcranial direct current stimulation (tDCS). Subjects will be compensated for their time.

DETAILED DESCRIPTION:
During the first study visit, subjects will receive a physical exam and an electroencephalogram (EEG), which measures brain activity. Research staff will put a cap on your head that has sensors which measure your brain activity. There is no risk of electrical shock. In addition to the sensors in the cap, two clips will be put on your ears. EEG activity will be collected for 20 minutes: you will have your eyes open for ten minutes, and then have your eyes closed for ten minutes.

Additional study visits will follow where we will perform five different procedures (neurofeedback, self-hypnosis, two levels of transcranial direct current stimulation, and meditation). All subjects will receive all five procedures and each procedure will be conducted for 20 minutes.

Self-Hypnosis Training: You will be given verbal suggestions from an audio recording (via headphones) for relaxation and changes in the way you think about pain.

Meditation: You will be asked to focus on a single word ("one") for the entire session.

Neurofeedback Training: During this procedure, three sensors will be placed on your scalp, and one on each earlobe. A small amount of electrode paste will be used when placing the sensor on your scalp. There is no risk of electrical shock. You will be able to see images on a computer screen that correspond to your brain waves. You will learn how to change your brainwaves by changing the images on the computer.

Electric Stimulation (two different levels): This procedure consists of direct stimulation of the brain by a weak electrical current. The two procedure sessions will differ in the characteristics of the stimulation. Two electrodes will be placed on your scalp and secured by a rubber strap. The tDCS procedure is considered experimental and is not currently approved by the FDA but has been studied previously, at the same level of current, in spinal cord injury.

Before and after each procedure we will complete a 10 minutes EEG assessment similar to what is described above. The final procedure session will end with a 20 minute assessment to determine how responsive you are to hypnosis. Each procedure visits may last up to three hours. There will be a total of 6 study visits over approximately 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Spinal Cord Injury
* 18 years of age or older
* Daily pain
* At least 12 months since injury
* Read speak and understand English

Exclusion Criteria:

* History of seizure disorder or non-normative brain activity
* Presence of traumatic brain injury or significant skull defects
* Exhibit moderate to severe cognitive impairment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects may be referred by their personal physician or enrolled after seeing recruitment flyers or brochures. Subjects will be recruited from a previous survey study conducted by the principal investigator, as well as a data registry maintained by the principal investigator. Individuals recruited from these studies were recruited primarily from rehabilitation clinics.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Current pain intensity after each study procedure will be the primary outcome measure. This pain intensity will be assessed using a 0 - 10 Numerical Rating Scale during the EEG (electroencephalogram) assessment after each intervention. | Ratings of current and of average, worst, and least pain intensity "during the past five minutes" will be obtained every 5 min during each of the EEG (electroencephalogram) assessments

SECONDARY OUTCOMES:
Study procedures will result in changes in the EEG (electroencephalogram) assessment. | Post procedure EEG (electroencephalogram) assessment is completed right after each study procedure
  Specifically these procedures will induce greater relative increases in alpha [7-12 Hz] bandwidth activity and greater relative decreases in beta (14-33 Hz) bandwidth activity, then either of the two control conditions.
The observed changes in EEG (electroencephalogram) bandwidth activity associated with these procedures will mediate the decreases in pain intensity. | Changes in the EEG (electroencephalogram) completed after each procedure will be related to the amount of pain relief experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Mark P. Jensen, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States